CLINICAL TRIAL: NCT06829069
Title: Knowledge, Attitude and Perception of Special Care Dentistry (SCD) Among Dental Students At the Faculty of Dentistry, Cairo University: a Cross-sectional Study
Brief Title: Knowledge, Attitude, and Perception of Special Care Dentistry (SCD) Among Dental Students At Cairo University.
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Gamal Fouad Mohamed Sherif, Doctor, Cairo University
Other Study IDs: CONS 2-2-1:Preventive measures
Record Dates: First submitted 2025-02-14; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Dental Health; Dental Education and Special Care Dentistry
Keywords: Special care dentistry; Dental education; Dental students; knowledge attitudes; Special needs patients; Oral health; Cross sectional study; Cairo University; Dental Curriculum; Egypt

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to understand dental students' perception of special needs dental care. The findings will offer analysis and valuable insights into students' interest, awareness and acceptance of Special Care Dentistry (SCD).The goal of this study is to identify gaps in dental education and training related to SCD. The results will help improve the curriculum and ensure that future dentists are better prepared to care for patients with special needs creating a more skilled and compassionate generation of professionals. This study is important because individuals with special needs often face challenges in accessing dental care, and improving dental education can help address this issue.

DETAILED DESCRIPTION:
Special Care Dentistry (SCD) is a specialized field dedicated to addressing the oral health needs of individuals with physical, mental, developmental, or cognitive impairments that make it challenging for them to access or receive standard dental care. These individuals are at a higher risk of oral diseases due to multiple barriers, including mobility restrictions, communication difficulties, behavioral challenges, and dependence on caregivers for oral hygiene maintenance. In addition to these personal and social barriers, the lack of adequate training among dental professionals further contributes to the difficulties special needs patients face in receiving proper dental care. According to the World Health Organization (WHO), over one billion people globally-approximately 15% of the population-live with disabilities. In Egypt, the 2017 census revealed that 10.77% of the population has some form of disability, with a significant number of adults aged 18-59 affected. Although Law No. 10 of 2018 on Persons with Disabilities emphasizes equal access to healthcare services, there is currently no structured national strategy that integrates SCD into the Egyptian healthcare system. While initiatives like the Takaful and Karama program provide financial and social support to individuals with disabilities, a dedicated framework for ensuring equitable access to dental care remains absent.Research has shown that individuals with special healthcare needs experience a higher prevalence of dental caries, periodontal disease, and other oral health issues due to challenges in maintaining oral hygiene and accessing dental services. Studies indicate that many dentists feel unprepared or reluctant to treat patients with disabilities, citing a lack of adequate training during their undergraduate education. In many dental schools, SCD is either insufficiently covered or entirely absent from the curriculum, leaving graduates without the necessary knowledge and clinical confidence to manage special needs patients effectively.Early exposure to SCD through structured theoretical education and hands-on clinical training has been shown to significantly improve dental students' competence and attitudes toward treating special needs patients. Countries such as Sweden, Denmark, Canada, and the United States have successfully integrated SCD into their dental education programs, ensuring that future dentists are equipped with the skills and knowledge required to provide inclusive oral healthcare. However, in Egypt, the extent to which dental students are trained in SCD remains unclear, highlighting the need for further investigation. This observational cross-sectional study aims to explore dental students' perceptions of SCD, focusing on their awareness, familiarity with SCD concepts, and attitudes toward managing patients with special healthcare needs. Additionally, it will assess students' evaluation of their current SCD education, identifying potential gaps that may hinder their preparedness to treat special needs patients in clinical practice. By analyzing these perspectives, the study seeks to provide valuable insights that can guide the development of more effective educational strategies. Enhancing dental education in this area is essential for producing a competent and confident workforce capable of addressing the unique oral healthcare needs of individuals with disabilities, ultimately improving access to equitable dental care.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled as a 4th, 5th, or 6th-year dental student
* Studying at the Faculty of Dentistry, Cairo University
* Willing to voluntarily participate in the study

Exclusion Criteria:

* Not enrolled in the 4th, 5th, or 6th year of the dental program at Cairo University
* Do not provide informed consent to participate
* Incomplete questionnaire responses

Ages: 20 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of undergraduate clinical dental students and interns from the Faculty of Dentistry, Cairo University. Participants will be drawn from 4th and 5th-year students and 6th-year interns to assess their perceptions, awareness, and preparedness regarding Special Care Dentistry (SCD). The study will use an electronic self-administered questionnaire to collect data over a 3-month period.
Sampling Method: Non-Probability Sample
Enrollment: 296 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Perception of dental students of Special Care Dentistry (SCD) regarding awareness, terminology and prior knowledge | Data would be collected online in the academic year 2024/2025
  Awareness, terminology and prior knowledge is measured by a validated questionnaire used in the study by (Ramadhani et al.2024)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty Of Dentistry, Cairo University, Cairo, Cairo Governorate, Egypt

REFERENCES:
- [Background] Ramadhani A, Izzati FR, Maharani DA, Malik NA, Setiawati F. Perception of Special-Care Dentistry among Dental Students at Universitas Indonesia: A Cross-Sectional Study. Dent J (Basel). 2024 Jan 22;12(1):19. doi: 10.3390/dj12010019. PMID 38275680